CLINICAL TRIAL: NCT04596566
Title: Can Personalized Diet Therapy Favourably Impact Disease Severity in Patients With Crohn's Disease
Brief Title: Modeling Patient Response to a Therapeutic Diet in Crohn's Disease
Acronym: TDI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Crohn's and Colitis Foundation (Other); University of Alberta (Other); University of Guelph (Other); University of British Columbia (Other); Alphabiomics (Unknown); University of Birmingham (Other)
Responsible Party: Principal Investigator, Maitreyi Raman, Clinical Associate Professor, Director Clinician Investigator Program (CIP), Medical Director Alberta's Collaboration of Excellence for Nutrition in Digestive Diseases (Ascend) , Medical Director Nutrition Services, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB19-0402
Record Dates: First submitted 2020-02-06; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CD-TDI (Other): Therapeutic diet Intervention ( CD-TDI )Group : Patients receiving CD-TDI will be offered patient-centered counseling for 12 weeks by a Registered Dietitian (RD) trained in the CD-TDI protocol with the goals of (a) identification and treatment of malnutrition if present, (b) targeted treatment of macro- and micronutrient deficiencies using whole foods;(c) increasing adherence to CD-TDI (d) multivitamin adherence and (e) reduced exposure to dietary antigens (e.g., maltodextrin, carrageenan, other food additives). They will receive a5 face-to-face appointment every 3 weeks with the study RD, and all other weekly appointments, which are 8 in number will be completed by phone.
  Interventions: Other: Therapeutic diet Intervention
- Conventional management (No Intervention): Conventional Management (Control) Group: CM patients will meet with the RD at baseline, week 7 and week 13 to complete their 24HR food recall twice on different days of the week, followed by a phone few days after the visit to complete the second part of the recall. They will be advised to follow their habitual diet and will be offered the dietary intervention at 14 weeks if they are still experiencing a disease flare

INTERVENTIONS:
Other: Therapeutic diet Intervention — The CD-TDI will incorporate global principles of the Mediterranean Diet (MD) refined to inform specific food choices based on our pilot data results and published literature reported mechanisms of mitigating inflammation in IBD. Patient compliance will be measured in three ways: 1) Mediterranean diet score checklists completed every 3 weeks at the face-to-face visits; 2) goal attainment scores captured weekly to identify the goals set, and the goals attained 47; and 3) fatty acids profiled from red blood cells to identify if fat intake reflects CD-TDI fat recommendations: 35% total calories from fat, 15% from MUFA, 13% from SFA and 6% from PUFA with a 8 n6:n:3 ratio of 8:1
  Arms: CD-TDI

SUMMARY:
BACKGROUND: There is an urgent need to understand the role of therapeutic dietary interventions on the treatment of inflammatory bowel disease (IBD). Although nutritional observational studies have examined associations between diet and the development of IBD, the relationship between dietary components and disease relapse is lacking. Despite the lack of a well-defined relationship between dietary determinants and disease relapse, patients with IBD frequently have a strong belief that diet has a key role in controlling the course of their disease, and maybe a trigger of disease relapse. This proposed randomized controlled trial (RCT) explores the efficacy of a Crohn's Disease (CD) Therapeutic Dietary Intervention (TDI) compared to conventional management (CM) to induce steroid-free clinical remission at week 13 in patients with active, mild-to-moderate luminal CD. For asymptomatic patients with active disease, efficacy of the diet will be explored by using fecal calprotectin and sonographic findings

Rationale: Our team of investigators recently compared a representative healthy population to patients with CD and identified CD patients have: lower intakes of polyunsaturated and monounsaturated fats and multiple micronutrients (vitamins C, D, thiamine magnesium, phosphorus, zinc, potassium), and; few patients with CD met criteria for an anti-inflammatory dietary pattern. Since the diet is a modifiable potential risk factor for disease recurrence in IBD, there is a strong rationale for the investigation of diet on disease course. Additionally, patients have expressed strong interest in identifying the relationships between diet and disease, therefore assigning priority to this theme is an opportunity to advance patient-oriented care.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary objectives

A) Symptomatic patients at the time of recruitment: Harvey Bradshaw Index (HBI) >5 to <16

1. To compare the proportion of patients in each study group at week 13 who are in corticosteroid-free (CF) clinical remission as measured by a Harvey Bradshaw Index (HBI) of <5 (primary endpoint)
2. To compare the proportion of patients in each study group at week 13 who are in biochemical remission as measured by a fecal calprotectin (FCP) of <250ug/g (primary endpoint).

B) Asymptomatic patients with active disease at the time of recruitment: Harvey Bradshaw Index (HBI) <5

1. To compare the proportion of patients in each study group at week 13 who are in biochemical remission as measured by a fecal calprotectin (FCP) of <250ug/g (primary endpoint).
2. To compare the proportion of patients in each study group at week 13 who are in clinical remission as measured by sonographic findings of inflammation (Bowel Wall thickening ≤ 3mm).

Secondary Hypothesis: The aim of the secondary objectives are to examine whether the dietary intervention has a significant effect on the gut microbiota and SCFAs in patients and whether this is associated with the intervention and disease recurrence at or before 13 weeks. The aim is also to examine whether the intervention has a significant effect on health-related quality of life.

* To identify the presence of within and between-group differences in microbial diversity, microbial composition, and abundance of short-chain fatty acids (SCFA) and SCFA-producing bacteria at baseline and 13weeks.
* To identify the presence of within and between-group differences in fecal SCFA concentrations at baseline and 13 weeks. To compare the proportion of patients in each study group at week14 that achieve clinical response (decrease in HBI>3points)

METHODS:

Randomized controlled trial design: This 3-year study, investigator-blinded, RCT (N=102) at the University of Calgary (UoC). Eligible participants will be randomly allocated in a 2:1 ratio to either the intervention group (CD-TDI) or conventional management (CM) alone (i.e., control group) for 13 weeks.

Conventional Management (Control) Group: CM patients will meet with the RD at baseline, week 7 and week 13 to complete their 24 hour food recall twice on different days of the week, followed by a phone few days after the visit to complete the second part of the recall. They will be advised to follow their habitual diet and will be offered the dietary intervention at 14 weeks if they are still experiencing a disease flare.

Therapeutic diet Intervention ( CD-TDI )Group : Patients receiving CD-TDI will be offered patient-centered counseling for 12 weeks by a Registered Dietitian (RD) trained in the CD-TDI protocol with the goals of (a) identification and treatment of malnutrition if present, (b) targeted treatment of macro- and micronutrient deficiencies using whole foods;(c) increasing adherence to CD-TDI (d) multivitamin adherence and (e) reduced exposure to dietary antigens (e.g., maltodextrin, carrageenan, other food additives). They will receive a5 face-to-face appointment every 3 weeks with the study RD, and all other weekly appointments, which are 8 in number will be completed by phone.

ELIGIBILITY:
Inclusion Criteria:

* (a)≥18 years;
* (b)diagnosis of mild-to-moderate luminal ileal, ileo-colonic or colonic CD
* (c) active disease with Harvey Bradshaw Index (HBI) <16 at time of recruitment;
* (d) for active symptomatic patients (HBI > 5 to <16) evidence of endoscopic disease activity within six months of enrolment (presence of ulceration ≥5mm ) and for active asymptomatic patients (HBI <5) sonographic findings of intestinal inflammation ≥3mm of bowel wall thickening)
* (e) biomarker evidence of inflammation fecal calprotectin at enrolment (FCP

  * 250microg/g).
* (f) < OR = 1 small bowel resection,
* (g) ability to provide informed consent

Exclusion Criteria:

* HBI >16 at time of recruitment;
* (b) fecal calprotectin < 250 microg/mg within 1 month prior to study enrollment;
* (c) patients with upper GI tract CD;
* (d) evidence of perianal or fistulizing disease; (
* e) >1 bowel surgery;
* (f) significant chronic disorders such as cardiac disease, renal failure, active pulmonary disease (these factors may influence dietary intake),
* (g) any psychiatric or neurocognitive comorbidity that would limit ability to follow an CD-TDI
* (h) laxative or antibiotics in the past 3 months and
* (i) presence of ostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-02-12 (Estimated); Study Completion 2023-06-12 (Estimated)

PRIMARY OUTCOMES:
Fecal calprotectin: Change is being assessed. | baseline, 7 and 13 weeks.
  <250 ug/mg with at least 100ug/g decline from baseline. FCP is a test used to detect inflammation in the colon and is associated with disease activity and severity.
Harvey Bradshaw Index (HBI): Change is being assessed | baseline, 7 and 13 weeks.
  HBI is a validated, non-invasive measure of disease activity captured through a symptom questionnaire and is a surrogate to endoscopic assessment to determine disease severity. HBI minimum value is "0" and maximum no limit. HBI < 5 is used in this study to indicate clinical remission. HBI> 16 means severe disease activity. Higher scores means worse outcomes. Based on experience with past recruitment for clinical trials, endoscopic assessment is not feasible due to access and patient acceptance.
Bowel wall thickness on sonographic findings and Fecal calprotectin: Change is being assessed. | baseline, 7 and 13 weeks for fecal calprotectin and baseline and week 13 for sonographic findings
  For asymptomatic patients with active disease at the time of recruitment (HBI <5 ) a combined primary endpoint using both FCP <250 ug/mg with at least 100ug/g decline from baseline and ultrasound findings of bowel wall thickening will be used.( ≤ 3mm).

SECONDARY OUTCOMES:
Fecal Microbiota Sequencing: change is being assessed. | baseline, 7 and 13 weeks
  Microbiome composition will be measured using shotgun metagenomic sequencing
Short chain fatty acids: Change is being assessed | baseline, 7 and 13 weeks
  Concentrations of fecal SCFA will be measured according to our previously published protocol. Fecal samples (150 mg) will be added to 1000 µL of 0.005 M aqueous sodium hydroxide containing internal standard (D3 caproic acid), and homogenized for 3 cycles using Fast Prep-24TM homogenizer (MP Biomedicals, Santa Anna, USA). The supernatant will be collected after centrifugation at 14,000 x g for 20 min. The derivatization using propyl chloroformate and analysis of the SCFAs using gas chromatography-mass spectrometry (GC-MS/MS) will be done as previously described
Health related quality of life: Change is being assessed. | baseline, 7 and 13 weeks
  Health-related quality of life will be measured using the 12-item short form-12. It comprises of two components physical health and mental Health. Scores range from 0 to 100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health.
Subjective global assessment: Change is being assessed | baseline, 7 and 13 weeks
  subjective global assessment is a validated tool to determine malnutrition status in patients with chronic disease. It is scored as A: Well-nourished; B: Mildly/moderately malnourished; C:Severely malnourished. "A" mean normal; "B" means some progressive nutritional loss; "C": means there is evidence of wasting and progressive symptoms
Dietary intake: Change is being assessed | baseline, 7 and 13 weeks
  Dietary intake and supplement use will be assessed at baseline (week 0),week 7 and week 13 using 2-24 Hour recalls using the multipass method.
Sedentary time: Change is being assessed | Baseline and week 13
  Sedentary time, will be assessed by the ActivPAL® inclinometer (PALTechnologies, Glasgow). ActivPAL® monitors are the most validated and widely used devices for measuring sitting, standing, and moving/stepping (and transitions in between). Inclinometers are small electronic devices worn discretely on the upper thigh. They measure duration and frequency of time spent sitting, standing and stepping (light ambulation), and number of postural changes. Materials: To capture all activities occurring throughout the day the ActivPAL® (captures lying, sitting, standing, and stepping).
CRP: Change is being assessed | Baseline and week 13
  C-reactive protein (mg/L)
Ferritin: Change is being assessed | Baseline and week 13
  Ferritin (Microgram/Litre)
Albumin: Change is being assessed | Baseline and week 13
  Albumin (g/L)
Vitamin D: Change is being assessed | Baseline and week 13
  Vitamins D (25OHD3) (nmol/L)
Cr: Change is being assessed | Baseline and week 13
  Creatinine( µmol/L)
Electrolytes: Change is being assessed | Baseline and week 13
  Electrolytes: Sodium (Na), potassium (K), chloride (Cl) mmol/L
Hb: Change is being assessed | Baseline and week 13
  Hemoglobin (Hb) (g/L)
Platelet: Change is being assessed | Baseline and week 13
  Platelet count (/L)
WBC: Change is being assessed | Baseline and week 13
  White blood cell count (WBC) (/L)

CONTACTS AND LOCATIONS:
Overall Officials: Maitreyi Raman, MD, Principal Investigator — University of Calgary
Locations (1):
- TRW building, Foothills, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers outside of the study team.

REFERENCES:
- [Derived] Haskey N, Letef C, Sousa JA, Yousuf M, Taylor LM, McKay DM, Ma C, Ghosh S, Gibson DL, Raman M. Exploring the connection between erythrocyte membrane fatty acid composition and oxidative stress in patients undergoing the Crohn's disease Therapeutic Diet Intervention (CD-TDI). Therap Adv Gastroenterol. 2025 Feb 16;18:17562848251314827. doi: 10.1177/17562848251314827. eCollection 2025. PMID 39963251
- [Derived] Raman M, Ma C, Taylor LM, Dieleman LA, Gkoutos GV, Vallance JK, McCoy KD, Lewis I, Jijon H, McKay DM, Mutch DM, Barkema HW, Gibson D, Rauch M, Ghosh S. Crohn's disease therapeutic dietary intervention (CD-TDI): study protocol for a randomised controlled trial. BMJ Open Gastroenterol. 2022 Jan;9(1):e000841. doi: 10.1136/bmjgast-2021-000841. PMID 35046093